CLINICAL TRIAL: NCT01511237
Title: PHPT-5 Second Phase: Perinatal Antiretroviral Intensification for the Prevention of Mother-to-child Transmission of HIV in Thai Women Having Received Less Than 8 Weeks of HAART During Pregnancy
Brief Title: Perinatal Antiretroviral Intensification for PMTCT of HIV in Late Comers
Acronym: PHPT-5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Harvard School of Public Health (HSPH) (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Marc Lallemant, Senior Researcher, Institut de Recherche pour le Developpement
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PHPT-5 Second Phase; R01HD052461 (NIH); R01HD056953 (NIH)
Record Dates: First submitted 2012-01-10; First posted 2012-01-18 (Estimated); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV-1 infection; Prophylaxis; Mother-to-child transmission HIV-1; Thailand; Developing Countries
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine; Zidovudine; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Perinatal intensification (Experimental): Perinatal antiretroviral intensification (study treatment):
  * Mothers: One NVP 200 mg tablet at onset of labor with continuation of HAART for four weeks postpartum
  * Newborn: AZT+3TC+ NVP for 2 weeks, followed by AZT+3TC for 2 weeks
  The standard of care in Thailand is defined as:
  * Maternal: ZDV 300 mg, 3TC 150mg and LPV/r 400/100 twice a day starting as soon possible after 14 weeks of pregnancy + ZDV 300 mg every 3 hours during labor
  * Newborn: ZDV 4 mg/kg every 12 hours for 4 weeks (ZDV dosing adjusted for premature infants).
  Interventions: Drug: Nevirapine, zidovudine, lamivudine

INTERVENTIONS:
Drug: Nevirapine, zidovudine, lamivudine — * Mothers: One NVP 200 mg tablet at onset of labor with continuation of HAART for four weeks postpartum
  * Newborn: AZT+3TC+ NVP for 2 weeks, followed by AZT+3TC for 2 weeks:
    * NVP syrup 2 mg/kg every 24 hours for seven days, followed by NVP syrup 4 mg/kg every 24 hours for seven days. Newborns less than 2500 g will be administered 2mg/kg NVP syrup at each intake
    * AZT syrup 4 mg/ kg will be given every 12 hours for four weeks (preterm infants less than 30 weeks will be administered 2 mg/kg every 12 hours; preterm 30-35 weeks will receive 2 mg/kg every 12 hours for the first 2 weeks, increased to 3 mg/kg for the next 2 weeks).
    * 3TC syrup 2 mg/kg every 12 hours for four weeks.

SUMMARY:
The purpose is to evaluate the efficacy of maternal and infant perinatal antiretroviral prophylaxis intensification for the prevention of mother-to-child intrapartum transmission of HIV-1 in women receiving less than 8 weeks of antiretroviral prophylaxis during pregnancy.

DETAILED DESCRIPTION:
Design: a multicenter, phase III, single-arm trial.

Perinatal antiretroviral intensification (study treatment) is defined as the addition to the standard of care* for mothers and infants of:

* Mothers: One NVP 200 mg tablet at onset of labor with continuation of HAART for four weeks postpartum
* Newborn: AZT+3TC+ NVP for 2 weeks, followed by AZT+3TC for 2 weeks:

  * NVP syrup 2 mg/kg every 24 hours for seven days, followed by NVP syrup 4 mg/kg every 24 hours for seven days. Newborns less than 2500 g will be administered 2mg/kg NVP syrup at each intake
  * AZT syrup 4 mg/ kg will be given every 12 hours for four weeks (preterm infants less than 30 weeks will be administered 2 mg/kg every 12 hours; preterm 30-35 weeks will receive 2 mg/kg every 12 hours for the first 2 weeks, increased to 3 mg/kg for the next 2 weeks).
  * 3TC syrup 2 mg/kg every 12 hours for four weeks.

    * The standard of care in Thailand is defined as:
* Maternal antiretroviral treatment: ZDV 300 mg, 3TC 150mg and LPV/r 400/100 twice a day starting as soon possible after 14 weeks of pregnancy + ZDV 300 mg every 3 hours during labor; this treatment may be continued, stopped or modified after delivery upon the recommendation of the internist.
* Newborn: ZDV 4 mg/kg every 12 hours for 4 weeks (ZDV dosing adjusted for premature infants).

ELIGIBILITY:
Eligibility. Pregnant women presenting at the prenatal clinics will be eligible if they are confirmed HIV-infected, intend to deliver and bring their infant to a study site for postnatal care for at least 6 months; at least 18 years old; and have given written informed consent to participate in the study, regardless of their CD4 cell count.

Maternal inclusion criteria:

* Evidence of HIV infection, as documented by two serology tests obtained at two different dates;
* All HIV infected pregnant women will be enrolled, either in the intervention arm or an observational study group.

  * Women more than 30 weeks gestational age at start of antiretroviral treatment will be eligible for the intervention. They will actually receive the study intervention if they present in labor after less than 8 weeks of treatment duration;
  * Women with no ANC will receive standard care and will be enrolled in an observational study group(and their infant will receive standard of care perinatal antiretroviral intensification)
  * Women with less than 30 weeks gestational age at start of treatment will receive standard care and will also be enrolled in the Observational Reference group;
* Agreement not to breastfeed;
* Consent to participate and to be followed for the duration of the study

Exclusion Criteria:

* Evidence of pre-existing fetal anomalies incompatible with life;
* Concurrent participation to any other clinical trial without prior agreement of the two study teams

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2011-12; Primary Completion 2015-06 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Rate of perinatal HIV transmission | 6 months
  HIV DNA PCR analysis at birth, 2 weeks, 1, 2, 4 and 6 months of age

SECONDARY OUTCOMES:
Safety for women and neonates | Up to 12 Months
  All grade 3 and 4 clinical adverse events and abnormal laboratory values in women will be recorded and graded according to the toxicity tables developed by the DAIDS
Pregnancy outcomes | Up to 12 Months
  Evaluation of the rates of live births and stillbirths, as well as birth weight, gestational age at delivery according to the results of the sonogram at first prenatal visit, newborn maturity (Ballard score).

CONTACTS AND LOCATIONS:
Overall Officials: Marc Lallemant, MD, Principal Investigator — Institut de Recherche pour le Developpement
Locations (36):
- Thailand (36):
  - Prapokklao Hospital, Chanthaburi, Changwat Chanthaburi
  - Mae Chan Hospital, Mae Chan, Changwat Chiang Rai
  - Phan Hospital, Phan, Changwat Chiang Rai
  - Banglamung Hospital, Bang Lamung, Changwat Chon Buri
  - Chonburi Hospital, Chon Buri, Changwat Chon Buri
  - Panasnikom Hospital, Chon Buri, Changwat Chon Buri
  - Chiang Kham Hospital, Chiang Kham, Changwat Phayao
  - Buddhachinaraj Hospital, Phitsanulok, Changwat Phitsanulok
  - Hat Yai Hospital, Hat Yai, Changwat Songkhla
  - Chomthong Hospital, Chom Thong, Chiang Mai
  - Fang Hospital, Fang, Chiang Mai
  - Nakornping Hospital, Mae Rim, Chiang Mai
  - Sanpatong Hospital, San Pa Tong, Chiang Mai
  - Chiangrai Prachanukroh Hospital, Chiang Rai, Chiangrai
  - Wiangpapao Hospital, Chiang Rai, Chiangrai
  - Chiang Saen Hospital, Chiang Saen, Chiangrai
  - Mahasarakam Hospital, Maha Sarakham, Mahasarakam
  - Nakhonpathom Hospital, Nakhon Pathom, Nakhonpathom
  - Samutprakarn Hospital, Mueang Samut Prakan, Samutprakarn
  - Samutsakhon Hospital, Samut Sakhon, Samutsakhon
  - Bhumibol Adulyadej Hospital, Bangkok
  - Nopparat Rajathanee Hospital, Bangkok
  - Bhuddasothorn Hospital, Chachoengsao
  - Health Promotion Center Region 10, Chiang Mai, Chiang Mai
  - Kalasin Hospital, Kalasin
  - Khon Kaen Hospital, Khon Kaen
  - Regional Health Promotion Centre 6, Khon Kaen, Khon Kaen
  - Lampang Hospital, Lampang
  - Lamphun Hospital, Lamphun
  - Maharaj Nakhon Si Thammarat Hospital, Nakhon Si Thammarat
  - Nong Khai Hospital, Nong Khai
  - Pranangklao Hospital, Nonthaburi
  - Phayao Provincial Hospital, Phayao
  - Vachira Phuket Hospital, Phuket
  - Rayong Hospital, Rayong
  - Songkhla Hospital, Songkhla

REFERENCES:
- [Background] Cressey TR, Punyawudho B, Le Coeur S, Jourdain G, Saenjum C, Capparelli EV, Jittayanun K, Phanomcheong S, Luvira A, Borkird T, Puangsombat A, Aarons L, Sukrakanchana PO, Urien S, Lallemant M; PHPT-5 study team. Assessment of Nevirapine Prophylactic and Therapeutic Dosing Regimens for Neonates. J Acquir Immune Defic Syndr. 2017 Aug 15;75(5):554-560. doi: 10.1097/QAI.0000000000001447. PMID 28489732
- [Result] Lallemant Marc, Amzal Billy, Urien Saik, Sripan Patumrat, Cressey Tim R, Ngo-Giang-Huong Nicole, Rawangban Boonsong, Sabsanong Prapan, Siriwachirachai Thitiporn, Jarupanich Tapnarong, Kanjanavikai Prateep, Wanasiri Phaiboon, Koetsawang Suporn, Jourdain Gonzague, Le Cœur Sophie, for the PHPT-5 team. 2015. -"Antiretroviral Intensification to Prevent Intrapartum HIV Transmission in Late Comers". 8th IAS Conference on HIV Pathogenesis Treatment & Prevention, Vancouver, Canada, 19-22 July 2015.
- [Result] Lallemant M, Amzal B, Sripan P, Urien S, Cressey TR, Ngo-Giang-Huong N, Klinbuayaem V, Rawangban B, Sabsanong P, Siriwachirachai T, Jarupanich T, Kanjanavikai P, Wanasiri P, Koetsawang S, Jourdain G, Le Coeur S; PHPT-5 site investigators. Perinatal Antiretroviral Intensification to Prevent Intrapartum HIV Transmission When Antenatal Antiretroviral Therapy Is Initiated Less Than 8 Weeks Before Delivery. J Acquir Immune Defic Syndr. 2020 Jul 1;84(3):313-322. doi: 10.1097/QAI.0000000000002350. PMID 32205720
- See also: PHPT-5 First Phase — http://www.clinicaltrials.gov/ct2/show/NCT00409591